CLINICAL TRIAL: NCT07388550
Title: Phase I Open-Label Safety Trial of Pembrolizumab for Neurological Post-Acute Sequelae of SARS-CoV-2 (PD1-PASC I)
Brief Title: Phase I Open-Label Safety Trial of Pembrolizumab for Neurological Post- Acute Sequelae of SARS-CoV-2 (PD1-PASC I)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002294; 002294-N
Record Dates: First submitted 2026-02-04; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: PASC; Long Covid; COVID; COVID-19; Postacute Sequelae of COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Single dose of Pembrolizumab 200 mg IV
  Interventions: Drug: Keytruda

INTERVENTIONS:
Drug: Keytruda — Single dose of Pembrolizumab 200 mg IV

SUMMARY:
Background:

SARS-CoV-2 is the virus that causes COVID-19. Some people who recover from an acute COVID-19 infection may continue to have symptoms that persist for months or years. These can include neurological symptoms, such as headaches, loss of taste or smell, dizziness, or trouble walking. Pembrolizumab is a drug approved to treat certain cancers. Researchers think this drug might reduce long-term neurologic symptoms after a COVID-19 infection.

Objective:

To test pembrolizumab in people with ongoing neurologic symptoms of COVID-19.

Eligibility:

People aged 18 years or older who had COVID-19 at least 6 months ago and have ongoing neurologic symptoms.

Design:

Participants will have 7 clinic visits in 7 months.

Participants will be screened. They will have a physical exam with blood tests. Swabs will be used to collect cells from inside the mouth and nose. They may opt to have an imaging scan.

Participants will also have other tests before they are given the study drug. These include eye and skin exams; tests of their memory and thinking; and tests of involuntary body functions, such as heart rate, blood pressure, sweating, and digestion. Their grip strength and walking pace will be measured. They will wear a heart rate monitor for 24 hours. They will wear devices on a wrist and thigh to measure activity for 10 days.

Participants will have a lumbar puncture (spinal tap): A thin needle will be inserted into their lower back to draw out a sample of the fluid around their spinal cord.

Pembrolizumab is given through a needle inserted into a vein. Participants will receive 1 dose of the drug.

Participants will have 4 follow-up visits over 6 months. Tests may be repeated during these visits.

DETAILED DESCRIPTION:
Study Description:

Despite clinical recovery from an acute SARS-CoV-2 infection, some individuals continue to experience ongoing symptoms for months to years afterwards, with many of these symptoms being neurologic. These neurologic post-acute sequelae of SARS-CoV-2 infection (Neuro-PASC) may be related to persisting viral antigen that leads to immune exhaustion. This study will primarily evaluate the safety of one dose of intravenous Pembrolizumab therapy in neuro-PASC participants with evidence of immune exhaustion. Pembrolizumab therapy may have positive clinical and laboratory effects on participants with persistent neurological symptoms, which will be measured as secondary outcomes.

Objectives:

Primary Objective:

-To determine the safety of a single dose of intravenous Pembrolizumab in participants with neurological postacute sequalae of SARS-CoV-2 infection.

Secondary objectives:

* To determine if one dose of intravenous Pembrolizumab can normalize markers of immune exhaustion in neuro-PASC.
* To determine if one dose of intravenous Pembrolizumab can lead to clinically relevant improvement in subjective and objective measures of ability.

Exploratory objectives:

* To determine if one dose of intravenous Pembrolizumab can change measures of SARS-CoV-2 antigen.
* To determine if one dose of intravenous Pembrolizumab can change measures of cytokines.
* To determine if one dose of intravenous Pembrolizumab can lead to improvement in subjective measures of symptoms.

Endpoints:

Primary endpoint:

- Number of adverse events and serious adverse events.

Secondary endpoints:

* Number of participants with normalization of PD-1 expression on CD8 T cells.
* Number of participants achieving a minimal clinically important difference in measures of function:

  * Work Disability Functional Assessment Battery (WDFAB)
  * PROMIS Global Health
  * Short Form 36 (SF-36)
  * PROMIS Cognitive Function
  * Montreal Cognitive Assessment (MoCA)
  * Incremental shuttle walk test

Exploratory endpoints:

* Detection of viral antigen
* Change in cytokine profile
* Statistically significant positive change from baseline:

  * PROMIS Depression score
  * PROMIS Anxiety
  * PROMIS Fatigue
  * PROMIS Sleep Disturbance
  * WHO post COVID-19 functional scale
  * Patient Post-COVID-19 Functional Status (PCFS) scale (0-4).
  * Provider Post-COVID-19 Functional Status (PCFS) scale (0-4).
  * FUNCAP55
  * Multidimensional Fatigue Inventory (MFI)
  * Pittsburgh Sleep Quality Index (PSQI)
  * Modified Depaul Symptom Questionnaire-Post Exertional Malaise (DSQ-PEM)
  * Post Exertional Malaise Visual Analogue Scale
  * Patient Global Impression of Change
  * Physician Global Impression of Change
  * Brief tablet-based neurocognitive testing
  * Near Infrared Spectroscopy of muscle
  * Actigraphy
  * Hand grip strength
  * Holter monitoring for 24 hrs
  * Orthostatic Intolerance Questionnaire/Orthostatic Intolerance Daily Activities Scale (OIQ/OIDAS)
  * Dysautonomia measures in response to the QSART, Valsalva maneuver or head-up tilt table testing.
  * Ophthalmology Examination

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged at least 18 or older.
* Provides documentation of at least one positive COVID-19 Test. Approved test can include the following:

  * PCR, NAA, or other EUA Approved test to confirm active COVID infection.
  * A positive anti-nucleocapsid antibody test.
  * A positive home Antigen test is acceptable when documentation of a photograph of the test with a phone-based date and time stamp is provided.
  * A positive anti-Spike antibody test is accepted in unvaccinated individuals or those who had antibody testing prior to vaccination.
* Previously diagnosed with mild-moderate COVID-19 (WHO Clinical Progression Scale between 2-5. Participants who had severe acute COVID-19 requiring hospitalization or ICU care are excluded.
* If participants had multiple SARS-CoV-2 infections, they would need to be at least 6 months after the last infection.
* All participants would need to have a negative SARS-CoV-2 nasal swab at the time of enrollment. Documentation of the SARS-CoV-2 infection that led to development of PASC confirmed either by a positive testing by a commercial laboratory or a positive home test followed by confirmatory nucleocapsid antibody testing.
* Exhibiting persistent neurologic symptoms evidenced by a self-reported illness narrative of the development of persistent PASC symptoms after recovering from a SARS-CoV-2 infection. These include symptoms such as fatigue, cognitive difficulties, sleep disturbances, orthostatic intolerance, and any ongoing issues with gait instability, vision, speech, swallowing, sensation, or strength. Symptoms must persist for at least 6 months after the diagnosis of acute COVID-19.
* All participants will have PD-1 expression on CD8 T cells that is one SD above the mean value of normal controls as established in the SINS Lab and published previously.
* Moderate to severe PASC symptom severity, as determined using PCFS (minimal score of 3).
* Ability of participant to understand and sign a written informed consent document.
* Prior completion of a clinical brain MRI after the diagnosis of COVID-19, or willingness to complete a brain MRI.
* Agrees not to have vaccinations over the course of the study.
* Participants of childbearing potential must agree to use a combination of contraception (defined as two forms of effective birth control) or have had surgical sterilization, from the time of enrollment until 4 months after the dose of study drug.
* Participants capable of sperm donation must agree to not donate sperm from the time of enrollment until 4 months after the dose of study drug.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* For participants who have not completed a brain MRI since onset of symptoms: inability to complete brain MRI with gadolinium including contraindicated metal in the body, prior allergic reaction to gadolinium, eGFR <45 mmol/L, or claustrophobia that is unable to be adequately treated with a low dose oral benzodiazepine.
* Contraindication to a research lumbar puncture, including use of anticoagulant medication, platelets < 50,000/uL, PT or PTT >1.5 x ULN for the NIH Clinical Center, if risk of lumbar puncture is increased for other reasons such as space occupying lesion, skin infection at site of the puncture or otherwise inability to complete the procedure.
* A condition that would significantly confound interpretation of the clinical and research tests as determined by the study investigators. This could include traumatic brain injury, substance use disorder, active malignancy, systemic immunologic disorders, current or previous long-term immune suppressive therapy.
* Any premorbid medical condition that would potentially cause fatigue and exercise intolerance. This includes many chronic medical diseases, such as congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, severe arthritis, uncontrolled asthma, renal failure, fibromyalgia, and ME/CFS.
* Symptom severity that makes it impossible for the participant to travel to NIH.
* Received a SARS-CoV-2 vaccine dose within less than 4 weeks of enrollment or is planning for any additional vaccines during the study.
* Prior treatment for PASC with immunomodulatory therapies such as check point inhibitors which in the opinion of the investigators could impact the outcome of this study.
* Current medications include oral steroids or other immunosuppressive medications which in the opinion of the investigators could impact the outcome of this study.
* Active participation in a clinical protocol which includes any intervention that may affect the results of the current study.
* Abnormal anti-thyroid panel (anti-TPO and anti-TG) test at screening visit.
* ANA titer of 1:80 or greater, positive anti-CCP.
* Abnormal screening blood tests exceeding any of the limits defined below or as deemed exclusionary by the investigators on review at baseline:

  * Aspartate aminotransferase and alanine aminotransferase values >2x upper limit of normal precluding the use of acetaminophen
  * Fasting triglyceride > 300 mg/dL.
  * Total bilirubin >2x upper limit of normal (unless participant has Gilbert syndrome)
  * Creatinine Clearance or eGFR <60 ml/minute (adjusted for race)
  * Hemoglobin < 10 g/dL
  * Absolute neutrophil count < 1000/microliter
  * Platelet count <130,000/mm3 (if platelet clumping is present on hematology slide review, platelet count <100,000/mm3 is considered exclusionary to study)
  * Hemoglobin A1c >= 6%
  * Thyroid-stimulating hormone (TSH) and adrenocorticotropic hormone (ACTH) within normal limits. If TSH is not within normal limits then the participant may be eligible if thyroxine (T4) is within normal limits. Participants are not excluded if they are on a stable dose of replacement thyroid medication; dose may be adjusted as needed.
* Previously documented anaphylaxis or severe systemic reaction to check point inhibitors, acetaminophen, or diphenhydramine.
* A severe psychiatric condition, which based on the assessment of the study investigators, will impact the ability to complete the study.
* Pregnancy or planning to get pregnant.
* Currently lactating/breastfeeding.
* Current or previous malignancy. A history of malignancy that has fully resolved with surgical resection only (e.g. no chemotherapy, radiation therapy, or immunotherapy) will be allowed.
* Current or past substance use disorder within last five years. Marijuana use within the past five years will not be an exclusion.
* Infection with HIV, tuberculosis, hepatitis B or C.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is to determine the safety of a single dose of intravenous Pembrolizumab in participants with neurological post-acute sequalae of SARS-CoV-2 infection. | From screening to Day 180.

SECONDARY OUTCOMES:
To determine if one dose of intravenous Pembrolizumab can lead to clinically relevant improvement in subjective and objective measures of ability. | Comparison between baseline, day 30, day 60 , and day 180 visits.
To determine if one dose of intravenous Pembrolizumab can normalize markers of immune exhaustion in neuro-PASC. | Comparison between baseline, day 30, day 60 , and day 180 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified subject data, harmonized to a common standard, are available to qualified researchers. Summary data are available to all. Data will be made available as soon as possible or at the time of associated publication. All data will be deposited in MapME/CFS (RTI).
Supporting Information: ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication.
Access Criteria: Request for data access will need to adhere to the standard processes per each repository. These repositories allow for querying and access to shared datasets.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002294-N.html